CLINICAL TRIAL: NCT02942875
Title: Motor Recovery of the Severely Impaired Paretic Upper Limb After Mirror Therapy in Sub-acute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, CHAN Wing Chiu, Doctoral research student, Department of Rehabilitation Science, Principal Investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20140613004
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Stroke
Keywords: upper limb; mirror therapy; rehabilitation; subacute
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirror therapy group (Experimental): MT group subjects will attend training sessions of bilateral upper limb exercise daily in the presence of the mirror.
  Interventions: Other: mirror therapy
- Control therapy group (Active Comparator): Control group subjects will undergo the same training sessions of bilateral upper limb exercise daily without mirror.
  Interventions: Other: control therapy

INTERVENTIONS:
Other: mirror therapy — During MT, subjects will sit in front of a table on which a mirror will be placed vertically in the space ipsilateral to the paretic upper limb with its reflective surface facing the unaffected upper limb. The subjects are required to look at the mirror to observe the reflective image of the unaffected arm from shoulder to the hand, while it is performing certain designated movements. At the same time, the affected arm will be required to follow the unaffected arm to practice the same movements.
  The upper limbs movements during the 30-min MT session are open and close of grasp; wrist flexion and extension; forearm supination and pronation; elbow flexion and extension; shoulder flexion and extension. A total of 120 repetitions for each action will be practiced.
  Arms: Mirror therapy group
Other: control therapy — Control group subjects undergo the same bilateral upper limbs exercise protocol without mirror
  Arms: Control therapy group

SUMMARY:
Our study aims at investigating the effect of intensive mirror therapy on the motor recovery of severely impaired paretic arm at subacute stroke.

DETAILED DESCRIPTION:
It was reported that upper limb hemiparesis happened in 80% of stroke patients and only 20% regained full arm function 6 months post stroke. The paretic upper arm accounted for 50% of the variance in functional limitation after stroke. Early and intensive upper limb intervention can promote motor recovery of paretic arm and is associated with better upper limb functional outcomes on 6 month post stroke. Mirror therapy (MT) is one of the potential approach in enhancing motor recovery of paretic arm after stroke. However, the effect of intensive MT on the motor recovery of severely impaired paretic arm after stroke has not been investigated. Knowledge on the effect of intensive MT on motor recovery can enhance formulation of effective and efficiency treatment protocol in stroke rehabilitation. Therefore, our study aims at investigating the effect of intensive MT on the motor recovery of severely impaired paretic arm of patients at subacute phase of stroke.

Stroke patients admitted to Haven of Hope Hospital will be screened according to inclusion and exclusion criteria. Eligible subjects will consent and be randomized into two groups: MT group- subjects will have daily two 30-min sessions of standardized bilateral upper limbs exercise with presence of mirror, 5 days per week for 4 consecutive weeks. During MT, a mirror is placed in the patient's mid-sagittal plane, with the reflecting surface facing the non-paretic upper limb so that the reflected image of this non-paretic limb would be perceived as the paretic upper limb. Subjects are instructed to watch at the movements of the reflected image of the non-paretic limbs and at the same time, the paretic upper limb should imitate the observed movements and be synchronized with those of the good side. Standardized bilateral upper limbs exercise (4 sets of 30 repetitions of shoulder, elbow, wrist and fingers movements) will be carried out within 30 min per session. Control group subjects will receive same daily two sessions of standardized bilateral upper limbs exercise without mirror, 5 days per week for 4 consecutive weeks. Motor functions of paretic arm of subjects measured by Fugl-Meyer Assessment (motor domain) and Wolf Motor Function Test will be assessed by independent assessor who is blinded to the group allocation of subjects before and after the 4-week intervention. Baseline comparison between the two groups was tested with independent t-test and the difference among and between groups after intervention will be tested by repeated measures ANOVA with level of significant at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* age 35 years or older
* first stroke within the first month after stroke onset;
* has upper limb paresis contralateral to the side of cerebral hemisphere with stroke;
* Presence of active movements (at least flicker of movement in gravity free position, but not able to accomplish full range of motion against gravity) at any one joint of shoulder, elbow and hand of hemiplegic arm, and Motricity Index less than 47.
* Able to follow instructions

Exclusion Criteria:

* has visual impairment not correctable by corrective lens;
* has cognitive impairment (Mini-Mental State Examination score < 22/30)
* has comprehension or expression aphasia;
* Presence of visuospatial neglect
* has premorbid neurological or musculoskeletal conditions that affect movements in the upper limbs

Ages: 35 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment arm score | 4 weeks

SECONDARY OUTCOMES:
Wolf Motor Function Test | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wing Chiu Chan, MSc, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Haven of Hope Hospital, Tseung Kwan O, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwakkel G, van Peppen R, Wagenaar RC, Wood Dauphinee S, Richards C, Ashburn A, Miller K, Lincoln N, Partridge C, Wellwood I, Langhorne P. Effects of augmented exercise therapy time after stroke: a meta-analysis. Stroke. 2004 Nov;35(11):2529-39. doi: 10.1161/01.STR.0000143153.76460.7d. Epub 2004 Oct 7. PMID 15472114
- [Background] Michielsen ME, Selles RW, van der Geest JN, Eckhardt M, Yavuzer G, Stam HJ, Smits M, Ribbers GM, Bussmann JB. Motor recovery and cortical reorganization after mirror therapy in chronic stroke patients: a phase II randomized controlled trial. Neurorehabil Neural Repair. 2011 Mar-Apr;25(3):223-33. doi: 10.1177/1545968310385127. Epub 2010 Nov 4. PMID 21051765
- [Result] Altschuler EL, Wisdom SB, Stone L, Foster C, Galasko D, Llewellyn DM, Ramachandran VS. Rehabilitation of hemiparesis after stroke with a mirror. Lancet. 1999 Jun 12;353(9169):2035-6. doi: 10.1016/s0140-6736(99)00920-4. No abstract available. PMID 10376620
- [Result] Barker WH, Mullooly JP. Stroke in a defined elderly population, 1967-1985. A less lethal and disabling but no less common disease. Stroke. 1997 Feb;28(2):284-90. doi: 10.1161/01.str.28.2.284. PMID 9040676
- [Result] Buccino G, Binkofski F, Fink GR, Fadiga L, Fogassi L, Gallese V, Seitz RJ, Zilles K, Rizzolatti G, Freund HJ. Action observation activates premotor and parietal areas in a somatotopic manner: an fMRI study. Eur J Neurosci. 2001 Jan;13(2):400-4. PMID 11168545
- [Result] Cacchio A, De Blasis E, De Blasis V, Santilli V, Spacca G. Mirror therapy in complex regional pain syndrome type 1 of the upper limb in stroke patients. Neurorehabil Neural Repair. 2009 Oct;23(8):792-9. doi: 10.1177/1545968309335977. Epub 2009 May 22. PMID 19465507
- [Result] Dohle C, Pullen J, Nakaten A, Kust J, Rietz C, Karbe H. Mirror therapy promotes recovery from severe hemiparesis: a randomized controlled trial. Neurorehabil Neural Repair. 2009 Mar-Apr;23(3):209-17. doi: 10.1177/1545968308324786. Epub 2008 Dec 12. PMID 19074686
- [Result] Ertelt D, Small S, Solodkin A, Dettmers C, McNamara A, Binkofski F, Buccino G. Action observation has a positive impact on rehabilitation of motor deficits after stroke. Neuroimage. 2007;36 Suppl 2:T164-73. doi: 10.1016/j.neuroimage.2007.03.043. Epub 2007 Mar 31. PMID 17499164
- [Result] Ezendam D, Bongers RM, Jannink MJ. Systematic review of the effectiveness of mirror therapy in upper extremity function. Disabil Rehabil. 2009;31(26):2135-49. doi: 10.3109/09638280902887768. PMID 19903124
- [Result] Feys H, De Weerdt W, Nuyens G, van de Winckel A, Selz B, Kiekens C. Predicting motor recovery of the upper limb after stroke rehabilitation: value of a clinical examination. Physiother Res Int. 2000;5(1):1-18. doi: 10.1002/pri.180. PMID 10785907
- [Result] Han C, Wang Q, Meng PP, Qi MZ. Effects of intensity of arm training on hemiplegic upper extremity motor recovery in stroke patients: a randomized controlled trial. Clin Rehabil. 2013 Jan;27(1):75-81. doi: 10.1177/0269215512447223. Epub 2012 Jul 16. PMID 22801472
- [Result] Hsieh YW, Wu CY, Liao WW, Lin KC, Wu KY, Lee CY. Effects of treatment intensity in upper limb robot-assisted therapy for chronic stroke: a pilot randomized controlled trial. Neurorehabil Neural Repair. 2011 Jul-Aug;25(6):503-11. doi: 10.1177/1545968310394871. Epub 2011 Mar 24. PMID 21436390
- [Result] Invernizzi M, Negrini S, Carda S, Lanzotti L, Cisari C, Baricich A. The value of adding mirror therapy for upper limb motor recovery of subacute stroke patients: a randomized controlled trial. Eur J Phys Rehabil Med. 2013 Jun;49(3):311-7. Epub 2013 Mar 13. PMID 23480975
- [Result] Kwakkel G, Kollen BJ, van der Grond J, Prevo AJ. Probability of regaining dexterity in the flaccid upper limb: impact of severity of paresis and time since onset in acute stroke. Stroke. 2003 Sep;34(9):2181-6. doi: 10.1161/01.STR.0000087172.16305.CD. Epub 2003 Aug 7. PMID 12907818
- [Result] Lamont K, Chin M, Kogan M. Mirror box therapy: seeing is believing. Explore (NY). 2011 Nov-Dec;7(6):369-72. doi: 10.1016/j.explore.2011.08.002. PMID 22051561
- [Result] Lee MM, Cho HY, Song CH. The mirror therapy program enhances upper-limb motor recovery and motor function in acute stroke patients. Am J Phys Med Rehabil. 2012 Aug;91(8):689-96, quiz 697-700. doi: 10.1097/PHM.0b013e31824fa86d. PMID 22469877
- [Result] Lin KC, Chuang LL, Wu CY, Hsieh YW, Chang WY. Responsiveness and validity of three dexterous function measures in stroke rehabilitation. J Rehabil Res Dev. 2010;47(6):563-71. doi: 10.1682/jrrd.2009.09.0155. PMID 20848369
- [Result] Rabadi MH, Rabadi FM. Comparison of the action research arm test and the Fugl-Meyer assessment as measures of upper-extremity motor weakness after stroke. Arch Phys Med Rehabil. 2006 Jul;87(7):962-6. doi: 10.1016/j.apmr.2006.02.036. PMID 16813784
- [Result] Mercier L, Audet T, Hebert R, Rochette A, Dubois MF. Impact of motor, cognitive, and perceptual disorders on ability to perform activities of daily living after stroke. Stroke. 2001 Nov;32(11):2602-8. doi: 10.1161/hs1101.098154. PMID 11692024
- [Result] Morris DM, Uswatte G, Crago JE, Cook EW 3rd, Taub E. The reliability of the wolf motor function test for assessing upper extremity function after stroke. Arch Phys Med Rehabil. 2001 Jun;82(6):750-5. doi: 10.1053/apmr.2001.23183. PMID 11387578
- [Result] Nakayama H, Jorgensen HS, Raaschou HO, Olsen TS. Recovery of upper extremity function in stroke patients: the Copenhagen Stroke Study. Arch Phys Med Rehabil. 1994 Apr;75(4):394-8. doi: 10.1016/0003-9993(94)90161-9. PMID 8172497
- [Result] Byl NN, Pitsch EA, Abrams GM. Functional outcomes can vary by dose: learning-based sensorimotor training for patients stable poststroke. Neurorehabil Neural Repair. 2008 Sep-Oct;22(5):494-504. doi: 10.1177/1545968308317431. PMID 18780884
- [Result] Ramachandran VS, Rogers-Ramachandran D, Cobb S. Touching the phantom limb. Nature. 1995 Oct 12;377(6549):489-90. doi: 10.1038/377489a0. No abstract available. PMID 7566144
- [Result] Thieme H, Mehrholz J, Pohl M, Behrens J, Dohle C. Mirror therapy for improving motor function after stroke. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD008449. doi: 10.1002/14651858.CD008449.pub2. PMID 22419334
- [Result] Thieme H, Bayn M, Wurg M, Zange C, Pohl M, Behrens J. Mirror therapy for patients with severe arm paresis after stroke--a randomized controlled trial. Clin Rehabil. 2013 Apr;27(4):314-24. doi: 10.1177/0269215512455651. Epub 2012 Sep 7. PMID 22960240
- [Result] Wolf SL, Catlin PA, Ellis M, Archer AL, Morgan B, Piacentino A. Assessing Wolf motor function test as outcome measure for research in patients after stroke. Stroke. 2001 Jul;32(7):1635-9. doi: 10.1161/01.str.32.7.1635. PMID 11441212
- [Result] Woodbury ML, Velozo CA, Richards LG, Duncan PW, Studenski S, Lai SM. Dimensionality and construct validity of the Fugl-Meyer Assessment of the upper extremity. Arch Phys Med Rehabil. 2007 Jun;88(6):715-23. doi: 10.1016/j.apmr.2007.02.036. PMID 17532892
- [Result] Wu CY, Huang PC, Chen YT, Lin KC, Yang HW. Effects of mirror therapy on motor and sensory recovery in chronic stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2013 Jun;94(6):1023-30. doi: 10.1016/j.apmr.2013.02.007. Epub 2013 Feb 15. PMID 23419791
- [Result] Yavuzer G, Selles R, Sezer N, Sutbeyaz S, Bussmann JB, Koseoglu F, Atay MB, Stam HJ. Mirror therapy improves hand function in subacute stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2008 Mar;89(3):393-8. doi: 10.1016/j.apmr.2007.08.162. PMID 18295613